CLINICAL TRIAL: NCT04212611
Title: Evaluation of Postoperative Analgesic Effects of Infraorbital Nerve Block by Levobupivacaine vs Ropivacaine After Cleft Palate Surgery: A Double-blinded Randomized Trial
Brief Title: Postoperative Analgesic Effects of Infraorbital Nerve Block in Cleft Palate Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences, Rishikesh (Other Government)
Responsible Party: Principal Investigator, ADABALA VIJAY BABU, Principal Investigator, All India Institute of Medical Sciences, Rishikesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12
Record Dates: First submitted 2019-12-19; First posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Experimental): Bilateral infra orbital blocks is performed using 2-3 mL of 0.375% levobupivacaine (group L)
  Interventions: Drug: INFRA ORBITAL BLOCK
- Group R (Experimental): Bilateral infra orbital blocks is performed using 2-3 mL of 0.375% ropivacaine (group R).
  Interventions: Drug: INFRA ORBITAL BLOCK

INTERVENTIONS:
Drug: INFRA ORBITAL BLOCK — Bilateral infra orbital blocks is performed using 2-3 mL of 0.375% levobupivacaine (group L) or ropivacaine (group R).
  Other Names: Group L and Group R

SUMMARY:
Cleft palate repair is a common surgery in children.. As such children with cleft palate tend to have a compromised airway due to associated congenital anomalies like Pierre Robin syndrome, Treacher Collins syndrome etc. After surgical correction of cleft palate, they are more prone to develop post-operative respiratory difficulty due to narrowed airway, increased secretion, pain and sedation caused by opioids.

Hence, regional block, using local anesthetics, becomes a good option in this surgery.

The supremacy of bilateral infraorital block using levo bupivacaine over intravenous fentanyl as well as over peri-incisional infiltration in has been shown .Levobupivacaine was developed after Ropivaciane was noted to be associated with less no of adverse events.. Ropivacaine has been used for peripheral block in children for surgical pain.

Though the use of Levobupivacaine in regional blocks in facial surgeries has been well established, studies are still needed to establish its supremacy over Ropivacaine in cleft palate surgeries

DETAILED DESCRIPTION:
When compared with ropivacaine, levobupivacaine is a newer, safer, longer acting local anesthetic with rapid onset and prolonged duration of analgesia and similar or more pronounced nerve blocking effects, depending on the concentration. Hence the present study is aimed to compare the effectiveness of 0.375% levobupivacaine and 0..375% ropivacaine in infra orbital block for cleft palate surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age of 2-12 years
* Children undergoing elective surgery for cleft palate.
* Children who are conscious and willing to participate in the study.
* Children who speak and understand English, Hindi, local or others.

Exclusion Criteria:

* Patient's refusal
* Allergy to the amide group of local anaesthetic agent
* Patient on anticoagulants or bleeding disorder
* Underlying other significant systemic diseases.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-20 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
change in the pain score from base line using the verbal rating scale (scale range: 0-5; 0: no pain, 5: strongest pain) on the day of surgery, as well as on the first and second postoperative days. | Till the second post operative day.
  Pain is measured using verbal rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Adabala, MD, Principal Investigator — AIIMS,Rishikesh
Locations (1):
- AIIMS Rishikesh, Rishikesh, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Yes
if study comes out with a positive result we will share the data with others
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: one year
Access Criteria: website